CLINICAL TRIAL: NCT04525833
Title: The Association of Liver Disease With Other Systemic Diseases, Focus on Diseases Progression, Treatments, and Clinical Outcomes: Analyses From the Hospital Database of Buddhist Tzu Chi Medical Foundation
Brief Title: Liver Disease and Other Systemic Diseases
Status: Recruiting | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Collaborators: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B10804008
Record Dates: First submitted 2020-08-04; First posted 2020-08-25 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Liver Diseases; Humans; Progression; Carcinogenesis; Fatty Liver Disease; Hepatitis C; Hepatitis B; Hepatocellular Carcinoma; Liver Cirrhoses; Treatment Outcome
MeSH Terms: conditions — Liver Diseases; Disease Progression; Carcinogenesis; Non-alcoholic Fatty Liver Disease; Hepatitis C; Hepatitis B; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Examine the association of chronic liver diseases (including hepatitis B, hepatitis C, alcoholic liver disease, fatty liver, liver cirrhosis, and hepatocellular carcinoma) with other systemic diseases by retrospectively analyzing the data from the Hospital Database of Buddhist Tzu Chi Medical Foundation.

DETAILED DESCRIPTION:
The global population is growing older over the next several decades. An essential component to keep people healthy, even with aging, is to prevent chronic disease progression and reduce associated complications. About 80% of older adults have one chronic condition, and 50% have at least two chronic disorders. Efforts to identify strategies to prevent or reduce the risk of chronic diseases and injuries and to widely apply effective interventions must be pursued. Because the liver is the largest solid organ in the human body with multiple functions, including nutrition, metabolism, proteins and biochemicals synthesis, and detoxification, its function is vital for the homeostasis of our body. The impairment of liver function may cause dysfunction or even shut down other systems in our body. Therefore, a better understanding of the pathogenesis of the liver disorder is not only a key issue in medical science, but it may also affect the general health and diseases of other body systems in a variety of ways. Finally, causing significant public health and economic losses globally. However, the impact and interactions of liver disorders on the progression, treatments, and prognosis of other systemic disorders, or vice versa, remain largely unknown. Recent studies have demonstrated the interactions between diabetes mellitus and liver diseases, and implying a possible deteriorating effect of diabetes on liver disease progression, treatment outcomes, and hepatic carcinogenesis. These lines of evidence not only verify the need for a better understanding of the interactions between liver and other disorders, but also justify a more extensive exploration of the interactions between liver diseases and other systemic disorders.

In this study, the investigators aim to examine the association of chronic liver diseases (including hepatitis B, hepatitis C, alcoholic liver disease, fatty liver, liver cirrhosis and hepatocellular carcinoma) with other systemic diseases by retrospectively analyzing the data from the Hospital Database of Buddhist Tzu Chi Medical Foundation. The investigators will examine the impacts of different systemic diseases on the disease progression and prognosis of Taiwanese patients with liver diseases and vice versa. Moreover, the investigators will also examine the different therapeutic strategies (including western, traditional Chinese medical, surgical or varied treatments) used for the treatments of liver diseases or systemic diseases, and their effects on the disease progression, long-term outcomes and prognosis of patients with chronic liver diseases or other systemic diseases in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who visited the gastroenterology clinics of the Tzu Chi Hospitals, Buddhist Tzu Chi Medical Foundation

Exclusion Criteria:

* Age younger than 18 or older than 99 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data collected from the Hospital Database of Buddhist Tzu Chi Medical Foundation
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of a new diagnosis of hepatocellular carcinoma (HCC) | From the date of enrollment until the date of first documented diagnosis of HCC, assessed up to 120 months.
  The new diagnosis of HCC is assessed every 3 months by abdominal sonography, and every 6 months with tumor markers (e.g. AFP), and confirmed by dynamic CT or MRI or pathological examination.
The incidence of a new diagnosis of any event of liver cirrhosis complications | From the date of enrollment until the date of first documented any event of liver cirrhosis complications, or date of death from any cause, whichever came first, assessed up to 120 months.
  Liver cirrhosis complications include ascites, esophageal or gastric varices bleeding, hepatorenal syndrome, spontaneous bacterial peritonitis, hepatic encephalopathy, hepatic pulmonary syndrome, liver failure (Child-Pugh score B or C), or liver transplant, that are assessed every 3 months clinically.
  A new diagnosis of any event of liver cirrhosis complications is a new documented any of the above liver cirrhosis complications, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Sheng Hsu, Ph.D, Principal Investigator — Liver Diseases Research Center, Taipei Tzu Chi Hospital
Locations (1):
- Ching-Sheng Hsu, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Wu CC, Tseng CW, Tseng KC, Chen YC, Wu TW, Chang SY, Chang YJ, Chao YC, Hsu CS. Radiofrequency ablation versus surgical resection for the treatment of solitary hepatocellular carcinoma 2 cm or smaller: A cohort study in Taiwan. J Formos Med Assoc. 2021 May;120(5):1249-1258. doi: 10.1016/j.jfma.2020.11.010. Epub 2020 Dec 4. PMID 33288401